CLINICAL TRIAL: NCT00103402
Title: A Randomized Clinical Trial to Evaluate the Efficacy and Safety of 10mg Alfuzosin in the Treatment of Chronic Prostatitis / Chronic Pelvic Pain Syndrome (CP/CPPS) in Recently-Diagnosed and/or Newly-Symptomatic Alpha-blocker Naïve Patients
Brief Title: Trial to Compare Alfuzosin Versus Placebo in the Treatment of Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPCRN2 Afluzosin; RFA-DK-03-004 (Other Grant/Funding Number: NIDDK); U01DK065209 (NIH)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Results first posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-05

CONDITIONS: Prostatitis
Keywords: Prostatitis; Non-bacterial Prostatitis; Prostatodynia; Alfuzosin; Alpha-adrenergic blocker
MeSH Terms: conditions — Prostatitis | interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alfuzosin (Experimental): 10 mg of alfuzosin once daily for 12 weeks
  Interventions: Drug: Alfuzosin
- Placebo (Placebo Comparator): 10 mg of an identical-looking placebo once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alfuzosin
  Arms: Alfuzosin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this randomized clinical trial is to evaluate the efficacy and safety of the alpha adrenergic blocker Alfuzosin (Uroxatral) in men with relatively new onset of chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS). Alfuzosin is a once daily (10 mg capsule), FDA approved medication for an indication in benign prostatic hyperplasia (BPH). The effectiveness of alfuzosin in improving lower urinary tract symptoms in patients with BPH has been documented in a number of placebo-controlled studies. A number of small studies have also suggested that alfuzosin ameliorates CP/CPPS symptoms through a similar alpha-blockade mechanism. This study will enable further testing of this hypothesis

DETAILED DESCRIPTION:
The two primary objectives of this study are:

* To compare 12 weeks of treatment with alfuzosin versus placebo in newly-diagnosed, alpha-blocker naive CP/CPPS participants with respect to the primary endpoint in the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI).
* To evaluate the safety and tolerability of 12 weeks of alfuzosin in newly-diagnosed, alpha-blocker naïve CP/CPPS participants.

The proportion of "responders" in each treatment arm will be compared to evaluate the overall safety and efficacy of alfuzosin as compared to placebo. Approximately 270 eligible patients, 135 per treatment arm, will be randomized and followed for a period of twelve (12) weeks after randomization.

There will be four research-clinic visits during which data for the primary and secondary outcome measures will be collected: visit 1 involves screening, visit 2 involves collection of baseline data and randomization, visit 3 is the 6-week evaluation, and visit 4 is the 12-week evaluation of the primary end point.

ELIGIBILITY:
Inclusion Criteria:

* Participant has signed and dated the appropriate Informed Consent document.
* Participant is male.
* Participant is at least 18 years of age.
* Participant has had symptoms of discomfort or pain in the pelvic region for at least a six-week interval at the time of presentation.
* Symptoms bothersome enough to prompt a physician visit have been present for two years or less.

Exclusion Criteria:

* Participant has evidence of facultative Gram negative or enterococcus with a value of greater than or equal to 1000 colony forming units (CFU) /ml in mid-stream urine (VB2).
* Participant has previously received alfuzosin (Uroxatral®), tamsulosin hydrochloride (Flomax®), doxazosin mesylate (Cardura®), terazosin hydrochloride (HCL) (Hytrin®), or other alpha-adrenergic receptor blockers for symptoms of CP/CPPS or within the past two years for any other reason.
* Participant has a history of prostate, penile, testicular, bladder, or urethral cancer or has undergone pelvic radiation, systemic chemotherapy, or intravesical chemotherapy.
* Participant has a history of moderate or severe hepatic impairment, severe renal sufficiency, severe or unstable cardiovascular (i.e. prolonged QT), respiratory, hematological, endocrinological, neurological or other somatic disorders.
* Participant has unilateral orchialgia without pelvic symptoms, active urethral stricture, or neurological disease or disorder affecting the bladder.
* Participant has uninvestigated, significant hematuria.
* Participant has undergone transurethral prostatectomy (TURP), transurethral incision of the prostate (TUIP), transurethral Incision or Resection of the Bladder Neck (TUIBN), transurethral microwave thermotherapy (TUMT), transurethral needle ablation (TUNA), balloon dilation of the prostate, open prostatectomy or any other prostate surgery or treatment such as cryotherapy or thermal therapy.
* Participant has a neurological impairment or psychiatric disorder preventing his understanding of consent and his ability to comply with the protocol.
* Participant is currently taking exclusionary medications such as potent CYP3A4 inhibitors (i.e. ketoconazole, itraconazole, or ritonavir) or erythromycin.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2005-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leroy Nyberg, MD PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); John Kusek, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (10):
- United States (9):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Northwestern U. Feinberg School of Medicine, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Harvard Medical School- Massachusetts General Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - University of Washington- Harborview Medical Center, Seattle, Washington
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data are available at the NIDDK Central Repository: https://repository.niddk.nih.gov/studies/cpcrn2-rct1/?query=CPCRN
URL: https://repository.niddk.nih.gov/studies/cpcrn2-rct1/?query=CPCRN

REFERENCES:
- [Background] Alexander RB, Propert KJ, Schaeffer AJ, Landis JR, Nickel JC, O'Leary MP, Pontari MA, McNaughton-Collins M, Shoskes DA, Comiter CV, Datta NS, Fowler JE Jr, Nadler RB, Zeitlin SI, Knauss JS, Wang Y, Kusek JW, Nyberg LM Jr, Litwin MS; Chronic Prostatitis Collaborative Research Network. Ciprofloxacin or tamsulosin in men with chronic prostatitis/chronic pelvic pain syndrome: a randomized, double-blind trial. Ann Intern Med. 2004 Oct 19;141(8):581-9. doi: 10.7326/0003-4819-141-8-200410190-00005. PMID 15492337
- [Background] Litwin MS. A review of the development and validation of the National Institutes of Health Chronic Prostatitis Symptom Index. Urology. 2002 Dec;60(6 Suppl):14-8; discussion 18-9. doi: 10.1016/s0090-4295(02)02296-3. PMID 12521581
- [Background] Schaeffer AJ; National Institute of Diabetes and Digestive and Kidney Diseases of the US National Institutes of Health. NIDDK-sponsored chronic prostatitis collaborative research network (CPCRN) 5-year data and treatment guidelines for bacterial prostatitis. Int J Antimicrob Agents. 2004 Sep;24 Suppl 1:S49-52. doi: 10.1016/j.ijantimicag.2004.02.009. PMID 15364307
- [Background] Schaeffer AJ, Landis JR, Knauss JS, Propert KJ, Alexander RB, Litwin MS, Nickel JC, O'Leary MP, Nadler RB, Pontari MA, Shoskes DA, Zeitlin SI, Fowler JE Jr, Mazurick CA, Kishel L, Kusek JW, Nyberg LM; Chronic Prostatitis Collaborative Research Network Group. Demographic and clinical characteristics of men with chronic prostatitis: the national institutes of health chronic prostatitis cohort study. J Urol. 2002 Aug;168(2):593-8. PMID 12131316
- [Background] Propert KJ, Alexander RB, Nickel JC, Kusek JW, Litwin MS, Landis JR, Nyberg LM, Schaeffer AJ; Chronic Prostatitis Collaborative Research Network. Design of a multicenter randomized clinical trial for chronic prostatitis/chronic pelvic pain syndrome. Urology. 2002 Jun;59(6):870-6. doi: 10.1016/s0090-4295(02)01601-1. PMID 12031372
- [Background] Schaeffer AJ, Datta NS, Fowler JE Jr, Krieger JN, Litwin MS, Nadler RB, Nickel JC, Pontari MA, Shoskes DA, Zeitlin SI, Hart C; Chronic Prostatitis Collaborative Research Network. Overview summary statement. Diagnosis and management of chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS). Urology. 2002 Dec;60(6 Suppl):1-4. doi: 10.1016/s0090-4295(02)01979-9. PMID 12521576
- [Result] Nickel JC, Krieger JN, McNaughton-Collins M, Anderson RU, Pontari M, Shoskes DA, Litwin MS, Alexander RB, White PC, Berger R, Nadler R, O'Leary M, Liong ML, Zeitlin S, Chuai S, Landis JR, Kusek JW, Nyberg LM, Schaeffer AJ; Chronic Prostatitis Collaborative Research Network. Alfuzosin and symptoms of chronic prostatitis-chronic pelvic pain syndrome. N Engl J Med. 2008 Dec 18;359(25):2663-73. doi: 10.1056/NEJMoa0803240. PMID 19092152

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alfuzosin | Placebo
Started | 138 | 134
Completed | 116 | 117
Not Completed | 22 | 17
Not completed — Adverse Event | 3 | 4
Not completed — Lost to Follow-up | 8 | 7
Not completed — Dissatisfied/No longer interested | 6 | 6
Not completed — Personal constraints/Other | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alfuzosin | Placebo | Total
Number analyzed (Participants) | 138 | 134 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.4) | 40.1 (12.3) | 40.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 138 | 134 | 272
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 14 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 16 | 36
  White | 88 | 97 | 185
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 7 | 24
NIH-CPSI [Mean (Standard Deviation); unit: units on a scale] — For the National Institutes of Health Chronic Prostatitis Symptom Index (NIHCPSI), higher scores indicate more severe symptoms (for the quality-of-life score, higher scores indicate a more negative effect). Score ranges are as follows: total score, 0 to 43; pain score, 0 to 21; urinary score, 0 to 10, quality-of-life score, 0 to 12; and average pain and urgency scores, 0 to 10.
  units on a scale
    Total score | 23.8 (6.3) | 25.1 (5.9) | 24.5 (6.1)
    Pain score | 11.1 (3.3) | 11.5 (3.4) | 11.3 (3.4)
    Urinary score | 4.5 (2.8) | 4.9 (2.9) | 4.7 (2.9)
    Quality of life score | 4.5 (1.1) | 4.7 (0.9) | 4.6 (1.0)
Likert Pain and Urgency Scale [Mean (Standard Deviation); unit: units on the scale] — For the Likert Pain and Urinary Urgency Scale, a score of 0 indicates no pain or urgency and a score of 10 indicates the most severe pain or urgency.
  units on the scale
    Average pain score | 4.9 (2.0) | 5.0 (1.9) | 5.0 (2.0)
    Urgency score | 4.4 (2.6) | 4.7 (2.6) | 4.6 (2.6)
McGill Pain Questionnaire [Mean (Standard Deviation); unit: units on a scale] — For the McGill Pain Questionnaire, higher scores indicate greater pain. Score ranges are as follows: total score, 0 to 45; sensory score, 0 to 33; affective score, 0 to 12. Population: Based on completed questionnaires
  units on a scale
    Total score: number analyzed (Participants) | 134 | 133 | 267
    Total score | 11.2 (8.6) | 11.6 (8.7) | 11.4 (8.7)
    Sensory score: number analyzed (Participants) | 134 | 133 | 267
    Sensory score | 8.6 (5.9) | 8.9 (6.2) | 8.8 (6.1)
    Affective score: number analyzed (Participants) | 134 | 133 | 267
    Affective score | 2.6 (3.3) | 2.6 (3.2) | 2.6 (3.3)
SF-12 [Mean (Standard Deviation); unit: units on a scale] — For the Medical Outcomes Study Short Form Health Survey 12 (SF-12), higher scores indicate better quality of life. Score range for both the physical and mental component summaries is 0 to 100. Population: Based on completed questionnaires
  units on a scale
    Physical component summary: number analyzed (Participants) | 136 | 130 | 266
    Physical component summary | 45.5 (9.6) | 45.6 (8.4) | 45.6 (9.0)
    Mental component summary: number analyzed (Participants) | 136 | 130 | 266
    Mental component summary | 44.0 (10.9) | 44.9 (10.2) | 44.5 (10.6)
Hospital Anxiety and Depression Scale [Mean (Standard Deviation); unit: units on a scale] — For the Hospital Anxiety and Depression Scale, higher scores indicate greater anxiety and depression; range, 0 to 42. Population: Based on completed questionnaires
  units on a scale
    number analyzed (Participants) | 137 | 133 | 270
    (all) | 12.8 (7.6) | 12.8 (7.1) | 12.8 (7.4)
International Index of Erectile Function [Mean (Standard Deviation); unit: units on a scale] — For the International Index of Erectile Function, higher scores indicate better sexual function; range, 0 to 75. Population: Based on completed questionnaires
  units on a scale
    number analyzed (Participants) | 133 | 126 | 259
    (all) | 53.5 (17.9) | 52.8 (17.4) | 53.2 (17.7)
Male Sexual Health Questionnaire [Mean (Standard Deviation); unit: units on a scale] — For the Male Sexual Health Questionnaire, higher scores indicate better function with respect to erection and ejaculation and greater satisfaction with sexual life; range, 0 to 40. Population: Based on completed questionnaires
  units on a scale
    number analyzed (Participants) | 130 | 126 | 256
    (all) | 30.0 (7.4) | 30.4 (6.6) | 30.2 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Decline in Total Score ≥4 for the NIH-CPSI Total Score From Baseline to 12 Weeks
Description: For the National Institutes of Health Chronic Prostatitis Symptom Index (NIHCPSI) total score, higher scores indicate more severe symptoms and scores range from 0 to 43. The primary outcome was a decline of at least 4 from baseline to 12 weeks
Time Frame: Baseline and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Alfuzosin | Placebo
Number analyzed (Participants) | 138 | 134
Participants | 68 | 66
Statistical Analysis 1: Comparison: Alfuzosin vs Placebo; Sample-size calculations were based on a 2-sided alpha of 0.05 with 80% power to detect a difference of 20 between response rates (40% placebo and 60% alfuzosin) for the Fisher's exact test. We calculated that a total sample of 270 participants would be required (135 per study group). This proposed sample size included a 20% increase to adjust for clustering within clinical sites and a 5% increase for interim monitoring; Test type: Superiority — The primary analysis compared rates for the primary outcome between study groups, using the exact conditional test version of the Mantel-Haenszel test to control for clustering by clinical center; p = 0.99, Mantel Haenszel; The exact conditional test version of the Mantel-Haenszel test was used to control for clustering by clinical center; Risk Difference (RD) = 0.1, 95% CI 2-sided [-11.2 to 11.0]

2. Secondary Outcome: Global Response Assessment (GRA)
Description: The response rate for the global response assessment was based on marked or moderate improvement at 12 weeks using a 7 point scale (marked worsening, moderate worsening, no change, slight improvement, moderate improvement, marked improvement).
Time Frame: 12 weeks
Population: The analysis population for this outcome is larger than the number of participants who completed the trial because a few participant answered this question without completing the other questionnaires
Measure: Count of Participants; unit: Participants
Arm/Group | Alfuzosin | Placebo
Number analyzed (Participants) | 119 | 123
Participants
  Marked improvement | 23 | 16
  Moderate improvement | 25 | 29
  Slight improvement | 26 | 32
  No change | 36 | 36
  Slight worsening | 6 | 5
  Moderate worsening | 2 | 4
  Marked worsening | 1 | 1
Statistical Analysis 1: Comparison: Alfuzosin vs Placebo; Marked or moderate improvement at 12 weeks Absolute Difference in Rates % (95% CI); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.90, Mantel Haenszel; Risk Difference (RD) = 1.8, 95% CI 2-sided [-9.0 to 2.5]

3. Secondary Outcome: Change in Subscales of the NIH-CPSI
Description: For the National Institutes of Health Chronic Prostatitis Symptom Index (NIHCPSI), higher scores indicate more severe symptoms (for the quality-of-life score, higher scores indicate a more negative effect). Score ranges are as follows: total score, 0 to 43; pain score, 0 to 21; urinary score, 0 to 10, quality-of-life score, 0 to 12; and average pain and urgency scores, 0 to 10.
Time Frame: Baseline and12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alfuzosin | Placebo
Number analyzed (Participants) | 116 | 117
units on a scale
  Total score | -7.1 (9.0) | -6.5 (8.5)
  Pain score | -3.3 (4.5) | -3.0 (4.4)
  Urinary score | -1.2 (2.6) | -1.0 (2.6)
  Quality-of-life score | -1.2 (1.5) | -1.2 (1.5)
Statistical Analysis 1: Comparison: Alfuzosin vs Placebo; Total score (0-43) change from baseline; Test type: Superiority; p = 0.70, t-test, 2 sided; Mean Difference (Net) = -0.5, 95% CI 2-sided [-2.7 to 1.5]
Statistical Analysis 2: Comparison: Alfuzosin vs Placebo; Pain score (0-21) change from baseline; Test type: Superiority; p = 0.64, t-test, 2 sided; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.4 to 0.8]
Statistical Analysis 3: Comparison: Alfuzosin vs Placebo; Urinary score (0-10) change from baseline; Test type: Superiority; p = 0.62, t-test, 2 sided; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.8 to 0.4]
Statistical Analysis 4: Comparison: Alfuzosin vs Placebo; Quality of life score (0-12) change from baseline; Test type: Superiority; p = .99, t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [-0.4 to 0.4]

4. Secondary Outcome: Change in Subscales of the McGill Pain Questionnaire
Description: For the McGill Pain Questionnaire, higher scores indicate greater pain. Score ranges are as follows: total score, 0 to 45; sensory score, 0 to 33; affective score, 0 to 12.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alfuzosin | Placebo
Number analyzed (Participants) | 112 | 116
units on a scale
  Total score | -3.4 (6.4) | -3.1 (6.5)
  Sensory score | -2.5 (5.0) | -2.3 (4.9)
  Affective score | -1.0 (2.1) | -0.9 (2.3)
Statistical Analysis 1: Comparison: Alfuzosin vs Placebo; McGill Total Score; Test type: Superiority; p = 0.45, t-test, 2 sided; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.8 to 1.2]
Statistical Analysis 2: Comparison: Alfuzosin vs Placebo; McGill Sensory Score; Test type: Superiority; p = 0.47, t-test, 2 sided; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.4 to 1.0]
Statistical Analysis 3: Comparison: Alfuzosin vs Placebo; McGill Affective Score; Test type: Superiority; p = 0.89, t-test, 2 sided; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.6 to 0.4]

5. Secondary Outcome: Change in Medical Outcomes Study Short Form 12
Description: For the Medical Outcomes Study Short Form Health Survey 12 (SF-12), higher scores indicate better quality of life. Score range for both the physical and mental component summaries is 0 to 100.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alfuzosin | Placebo
Number analyzed (Participants) | 115 | 113
units on a scale
  Physical component | 3.0 (7.4) | 3.5 (8.1)
  Mental component | 4.0 (10.5) | 1.9 (10.6)
Statistical Analysis 1: Comparison: Alfuzosin vs Placebo; Physical component summary (0-100) change in scores; Test type: Superiority; p = 0.60, t-test, 2 sided; Mean Difference (Net) = -0.5, 95% CI 2-sided [-2.3 to 1.3]
Statistical Analysis 2: Comparison: Alfuzosin vs Placebo; Mental component summary (0-100) Absolute Difference between Groups (95% CI); Test type: Superiority; p = 0.16, t-test, 2 sided; Mean Difference (Net) = 2.1, 95% CI 2-sided [-0.4 to 4.6]

6. Secondary Outcome: Change in Hospital Anxiety and Depression Scale
Description: For the Hospital Anxiety and Depression Scale, higher scores indicate greater anxiety and depression; range, 0 to 42.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alfuzosin | Placebo
Number analyzed (Participants) | 115 | 117
units on a scale | -2.6 (5.7) | -1.5 (5.5)
Statistical Analysis 1: Comparison: Alfuzosin vs Placebo; Test type: Superiority; p = 0.08, t-test, 2 sided; Mean Difference (Net) = -1.1, 95% CI 2-sided [-2.4 to 0.2]

7. Secondary Outcome: Change in International Index of Erectile Dysfunction (IIEF)
Description: For the International Index of Erectile Function, higher scores indicate better sexual function; range, 0 to 75.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alfuzosin | Placebo
Number analyzed (Participants) | 110 | 109
units on a scale | 0.5 (12.7) | -0.2 (14.7)
Statistical Analysis 1: Comparison: Alfuzosin vs Placebo; Test type: Superiority; p = 0.94, t-test, 2 sided; Risk Difference (RD) = 0.7, 95% CI 2-sided [-2.6 to 4.0]

8. Secondary Outcome: Change in Male Sexual Health Questionnaire
Description: For the Male Sexual Health Questionnaire, higher scores indicate better function with respect to erection and ejaculation and greater satisfaction with sexual life; range, 0 to 40.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alfuzosin | Placebo
Number analyzed (Participants) | 107 | 111
units on a scale | 1.7 (4.5) | 0.6 (6.8)
Statistical Analysis 1: Comparison: Alfuzosin vs Placebo; Test type: Superiority; p = 0.06, t-test, 2 sided; Mean Difference (Net) = 1.1, 95% CI 2-sided [-0.3 to 2.5]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Alfuzosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/134
Serious Adverse Events (participants affected / at risk) | 1/138 | 2/134
Other Adverse Events (participants affected / at risk) | 40/138 | 46/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alfuzosin (N=138) | Placebo (N=134)
Spontaneous pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Traumatic head laceration (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alfuzosin (N=138) | Placebo (N=134)
Constitutional events (General disorders) | 4 (4) | 7 (7)
Gastrointestinal events (Gastrointestinal disorders) | 10 (10) | 13 (13)
Neurologic events (Nervous system disorders) | 11 (11) | 6 (6)
Pain in any body system (General disorders) | 15 (15) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No